CLINICAL TRIAL: NCT06557811
Title: Effect of Oral Semaglutide on Epicardial and Pericoronary Adipose Tissues in Type 2 Diabetes After Myocardial Infarction: a Randomized and Double-blind Clinical Trial
Brief Title: Effect of Oral Semaglutide on Epicardial and Pericoronary Adipose Tissues in Type 2 Diabetes After Myocardial Infarction
Acronym: SemaFatCard
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Jr, Professor Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 75667623.1.0000.0068
Record Dates: First submitted 2024-08-06; First posted 2024-08-16 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Patients; Acute Myocardial Infarction
Keywords: Diabetes; Acute myocardial infarction; Oral Semaglutide
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Diabetic patients who suffered acute myocardial infarction will be divided into 2 groups, an arm that will receive medication and another arm placebo (control population).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind, meaning both the research participants and the outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Other): 2 groups: This group will receive semaglutide
  Interventions: Drug: Semaglutide
- Placebo (Other): 2 groups: This group will receive placebo (control population).
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — After randomization, each patient will receive four blisters of 3 mg tablets (semaglutide or placebo) and four blisters of 7 mg tablets (semaglutide or placebo), to be taken before breakfast. After 60 days, the patient will receive a 14 mg dose (a total of 16 blisters with 7 tablets each). The possibility of maintaining the 14 mg dose of the study drug or reducing it to 7 mg will be evaluated depending on side effects and tolerability.
  Other Names: Rybelsus

SUMMARY:
The goal of this clinical trial is to investigate the ability of oral semaglutide to reduce pericardial and perivascular fat as well as coronary plaque in type 2 diabetic patients after acute myocardial infarction. Patients of both sexes, aged 50 years or older, diagnosed with type 2 diabetes and with a previous acute myocardial infarction between more than 2 and less than 9 months ago, will be included.

The primary objective is to investigate the ability of oral semaglutide to reduce pericardial and perivascular fat in type 2 diabetics after myocardial infarction.

The primary outcome will be composed of three measures:

Measurement of pericardial adipose tissue at 180 days; Measurement of the perivascular adipose tissue attenuation index at 180 days; Measurement of the fat attenuation index at 180 days.

To assess the degree of epicardial and perivascular fat attenuation, coronary artery computed tomography will be performed, and to evaluate the left ventricular ejection fraction, transthoracic echocardiography will be conducted.

Oral semaglutide may reduce pericardial and/or perivascular fat in diabetics after acute myocardial infarction.

DETAILED DESCRIPTION:
TITLE: Effect of Oral Semaglutide on Epicardial and Pericoronary Adipose Tissues in Type 2 Diabetic Patients After Myocardial Infarction.

OBJECTIVE: This randomized, placebo-controlled study primarily aims to demonstrate the effect of oral semaglutide on pericardial and pericoronary adipose tissues, atherosclerotic plaque, and the vascular lumen in patients with T2D after myocardial infarction through CCT and CTA analysis, with a secondary objective of analyzing anthropometric markers, cardiac markers, and insulin resistance.

MATERIAL AND METHODS: Equipment: Cardiac Computed Tomography (CCT) and Echocardiography: A standard CTA protocol using a 320 detector-row scanner (Aquillion ONE, Canon Medical Systems, Ottawa, Japan), including coronary calcium score (CCS) and CTA, will be performed. To achieve a heart rate < 65 bpm during acquisition, patients will receive oral metoprolol (50-100 mg) or intravenous metoprolol (up to 15 mg in 5 mg increments). Fast-acting sublingual nitrate (2.5-5 mg) will also be administered to all patients before scanning. After CCS acquisition, ECG-triggered CTA will be performed with 70 mL of non-ionic contrast (Iopromide 370 mg iodine/mL, Bayer Schering Pharma, Berlin, Germany), injected intravenously at 5.0 mL/s, followed by 30-40 mL of saline. The CTA parameters are as follows: collimation 0.5 mm, rotation time 400 ms, tube voltage and current 100-120 kV and 250-550 mA, adjusted to body mass index. To be performed during Visits 1 and 2:

* Coronary Computed Tomography Angiography (CTA) in the proximal segment of the right coronary artery and/or anterior descending coronary artery.
* Cardiac Markers: Troponin I, CK-MB, C-Reactive Protein, Interleukin 6.
* Metabolic Markers: Measurement of neck circumference, hepatic steatosis (Abdominal Ultrasound), Fasting Glycemia, HbA1c, Basal Insulin and HOMA-IR, Cystatin C, Total Cholesterol and Fractions, Uric Acid, TSH and Free T4.
* Anthropometric and Clinical Markers: Body Weight, Body Mass Index (BMI) = weight / height², Abdominal Waist (AW), AW/Height Ratio, Blood Pressure, and Heart Rate.

STUDY DESIGN: Prospective, placebo-controlled, double-blind, single-center randomized study with 4 phases: First phase: Screening of chronic patients who had AMI with T2D for more than 1 month and less than 6 months in the InCor database, according to inclusion criteria. The patient will be called for Visit 1 (inclusion). If the screening is successful, the patient will be fully informed about this study and will read and freely sign the Informed Consent Form (ICF). After this, a clinical consultation will be conducted, anthropometric data, blood pressure, and heart rate will be measured, and the exams of CCT, CTA, Abdominal Ultrasound, Echocardiography, and other markers described will be ordered to enter the 1st phase of the study and receive randomized oral semaglutide/placebo treatment on the day of Visit 1. Randomization: The start of randomization will be considered as day one. The other phases will be counted from the start of randomization. Phone calls during the 2nd and 3rd phases will ask the following questions: 1) Is the patient using the medication correctly? If not, the patient will be invited for an extra visit. 2) Is the patient experiencing any Adverse Events (AE)? If yes, the patient will be invited for an extra visit. 4th Phase (Visit 2): It will be asked if the patient used the medication/placebo correctly, if any AE occurred, a clinical consultation will be conducted, and the exams of CCT, CTA, Abdominal Ultrasound, Echocardiography, and other described markers will be ordered.

STATISTICAL ANALYSIS: Qualitative characteristics will be described according to the groups using absolute and relative frequencies, and the association between groups will be verified at Visit 1 using chi-square tests or exact tests. Quantitative characteristics will be described according to the groups using summary measures (mean, standard deviation, median, minimum, and maximum) and compared at baseline using Student's t-test or Mann-Whitney tests according to the probability distribution of the data. The characteristics of interest will be described according to the groups throughout the follow-up using summary measures and compared between groups and evaluation moments using generalized estimation equations with appropriate distributions and linkages, followed by Bonferroni multiple comparisons when necessary. IBM-SPSS for Windows version 22.0 software will be used for the analysis, and Microsoft Excel 2010 software will be used for data tabulation. Tests will be performed with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

Male or female patient aged 50 years or older at the time of screening, diagnosed with type 2 diabetes and with a previous acute myocardial infarction more than 2 and less than 9 months ago, with the following conditions:

1. Signed Informed Consent Form.
2. BMI ≥ 25 and < 40 kg/m².
3. The following glucose-lowering agents are permitted: any insulin, insulin analogs, sulfonylureas, meglitinides, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, and SGLT-2 inhibitors (iSGLT2).
4. Patients using iSGLT2 will not be excluded because they receive this medication at no cost at InCor with benefits for the treatment of type 2 diabetes. Furthermore, there would be an impact on ethical issues and the control of this prescription in other clinics. Thus, we will list the patients using SGLT2 inhibitors and statistically evaluate the comparison with the group that did not use this medication.

Exclusion Criteria:

1. Patients with type 1 diabetes.
2. Type 2 diabetes currently or previously treated (within 90 days prior to screening) with any GLP-1RA and DPP-4 inhibitor.
3. Those not properly treated for previously diagnosed hypothyroidism.
4. Diagnosed with NYHA class IV heart failure.
5. Myocardial infarction more than 9 months after diagnosis.
6. Any of the following: myocardial infarction, stroke, or hospitalization for unstable angina or transient ischemic attack within 60 days before screening.
7. Any contraindication present in the package insert for the use of GLP1-RA or Oral Semaglutide.
8. Desire to become pregnant.
9. Previous history of pancreatitis (acute or chronic).
10. Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
11. History of major surgical procedures involving the stomach, potentially affecting the absorption of the test product (e.g., subtotal and total gastrectomy, vertical gastrectomy, gastric bypass surgery).
12. Planned and known coronary, carotid, or peripheral arterial revascularization on the day of screening.
13. Chronic or intermittent hemodialysis, peritoneal dialysis, or severe renal insufficiency (corresponding to eGFR < 30 mL/min/1.73 m²) - due to CT specifications reported below.

    History or presence of malignant neoplasm in the last 5 years (except basal cell and squamous cell skin cancer and carcinoma in situ).
14. History of diabetic ketoacidosis.
15. Participation in another clinical trial investigating a drug.
16. Participation in a clinical trial specifically evaluating stent(s) will be allowed.
17. Uncontrolled systemic arterial hypertension with multiple antihypertensive agents.
18. Any disorder that, in the opinion of the researcher, may compromise patient safety or protocol compliance.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of pericardial adipose tissue at 180 days | 180 days
  Measurement of pericardial adipose tissue (cm³)
Measurement of the fat attenuation index at 180 days | 180 days
  Measurement of the fat attenuation index (Hounsfield units (HU))
Measurement of the perivascular adipose tissue attenuation index at 180 days | 180 days
  Measurement of the perivascular adipose tissue attenuation index (Hounsfield units (HU))

SECONDARY OUTCOMES:
Determination of metabolic marker levels fasting blood glucose | 180 days
  Determination of metabolic marker level: fasting blood glucose (mg/dL)
Determination of metabolic marker levels HbA1c | 180 days
  Determination of metabolic marker level: HbA1c (%)
Determination of metabolic marker levels Insulin | 180 days
  Determination of metabolic marker level: Insulin (µU/mL)
Determination of metabolic marker levels HOMA-IR | 180 days
  Determination of metabolic marker level:HOMA-IR
Determination of metabolic marker levels total cholesterol and fractions | 180 days
  Determination of metabolic marker levels:total cholesterol and fractions (mg/dL)
Determination of metabolic marker levels uric acid | 180 days
  Determination of metabolic marker levels:uric acid (mg/dL)
Determination of metabolic marker levels TSH | 180 days
  Determination of metabolic marker levels:TSH (µUI/mL)
Determination of metabolic marker levels free T4 | 180 days
  Determination of metabolic marker levels: free T4 (ng/dL)
Determination of complete blood count with platelet count | 180 days
  Determination of complete blood count: Hemoglobin (g/dL)
Determination of complete blood count | 180 days
  Determination of complete blood count: Hematocrit (%)
Determination of platelet count | 180 days
  Determination of platelet count (x10^3/µL)
Determination of cardiac marker levels Troponin I | 180 days
  Measure of cardiac marker level: Troponin I (ng/mL)
Determination of cardiac marker levels CK-MB | 180 days
  Measure of cardiac marker level: CK-MB (ng/mL)
Determination of cardiac marker levels C-Reactive Protein | 180 days
  Measure of cardiac marker level: C-Reactive Protein (mg/L)
Determination of cardiac marker levels Interleukin 6 | 180 days
  Measure of cardiac marker level:Interleukin 6 (pg/mL)
Determination of cardiac marker levels NT-proBNP | 180 days
  Measure of cardiac marker level: NT-proBNP (pg/mL)
Determination of anthropometric measurements body mass index | 180 days
  Determination of anthropometric measurement: body mass index (kg/m2)
Determination of anthropometric measurements Neck Circumference | 180 days
  Determination of anthropometric measurement: Neck Circumference (cm)
Determination of anthropometric measurements Body Weight | 180 days
  Determination of anthropometric measurement: Body Weight (kg)
Determination of anthropometric measurements Abdominal Waist | 180 days
  Determination of anthropometric measurement: Abdominal Waist (cm)
Determination of anthropometric measurements Waist-to-Height Ratio | 180 days
  Determination of anthropometric measurement:Waist-to-Height Ratio
Determination of anthropometric measurements Blood Pressure | 180 days
  Determination of anthropometric measurement: Blood Pressure (mmHg)
Determination of anthropometric measurements Heart Rate | 180 days
  Determination of anthropometric measurement:Heart Rate (bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos V Serrano Junior, MD PHD, Principal Investigator — InCOR- University of Sao Paulo
Locations (1):
- ARO (Academic Research Organization), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Tsaban G, Wolak A, Avni-Hassid H, Gepner Y, Shelef I, Henkin Y, Schwarzfuchs D, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Tene L, Zelicha H, Yaskolka-Meir A, Komy O, Bilitzky A, Chassidim Y, Ceglarek U, Stumvoll M, Bluher M, Thiery J, Dicker D, Rudich A, Stampfer MJ, Shai I. Dynamics of intrapericardial and extrapericardial fat tissues during long-term, dietary-induced, moderate weight loss. Am J Clin Nutr. 2017 Oct;106(4):984-995. doi: 10.3945/ajcn.117.157115. Epub 2017 Aug 16. PMID 28814394
- [Background] Iacobellis G. Epicardial adipose tissue in endocrine and metabolic diseases. Endocrine. 2014 May;46(1):8-15. doi: 10.1007/s12020-013-0099-4. Epub 2013 Nov 23. PMID 24272604
- [Background] Lazaros G, Antonopoulos A, Antoniades C, Tousoulis D. The Role of Epicardial Fat in Pericardial Diseases. Curr Cardiol Rep. 2018 Apr 19;20(6):40. doi: 10.1007/s11886-018-0986-7. PMID 29675684
- [Background] Russo R, Di Iorio B, Di Lullo L, Russo D. Epicardial adipose tissue: new parameter for cardiovascular risk assessment in high risk populations. J Nephrol. 2018 Dec;31(6):847-853. doi: 10.1007/s40620-018-0491-5. Epub 2018 Apr 27. PMID 29704210
- [Background] Nagy E, Jermendy AL, Merkely B, Maurovich-Horvat P. Clinical importance of epicardial adipose tissue. Arch Med Sci. 2017 Jun;13(4):864-874. doi: 10.5114/aoms.2016.63259. Epub 2016 Oct 26. PMID 28721155
- [Background] Horckmans M, Bianchini M, Santovito D, Megens RTA, Springael JY, Negri I, Vacca M, Di Eusanio M, Moschetta A, Weber C, Duchene J, Steffens S. Pericardial Adipose Tissue Regulates Granulopoiesis, Fibrosis, and Cardiac Function After Myocardial Infarction. Circulation. 2018 Feb 27;137(9):948-960. doi: 10.1161/CIRCULATIONAHA.117.028833. Epub 2017 Nov 22. PMID 29167227
- [Background] Young LH, Viscoli CM, Curtis JP, Inzucchi SE, Schwartz GG, Lovejoy AM, Furie KL, Gorman MJ, Conwit R, Abbott JD, Jacoby DL, Kolansky DM, Pfau SE, Ling FS, Kernan WN; IRIS Investigators. Cardiac Outcomes After Ischemic Stroke or Transient Ischemic Attack: Effects of Pioglitazone in Patients With Insulin Resistance Without Diabetes Mellitus. Circulation. 2017 May 16;135(20):1882-1893. doi: 10.1161/CIRCULATIONAHA.116.024863. Epub 2017 Feb 28. PMID 28246237
- [Background] Kernan WN, Viscoli CM, Furie KL, Young LH, Inzucchi SE, Gorman M, Guarino PD, Lovejoy AM, Peduzzi PN, Conwit R, Brass LM, Schwartz GG, Adams HP Jr, Berger L, Carolei A, Clark W, Coull B, Ford GA, Kleindorfer D, O'Leary JR, Parsons MW, Ringleb P, Sen S, Spence JD, Tanne D, Wang D, Winder TR; IRIS Trial Investigators. Pioglitazone after Ischemic Stroke or Transient Ischemic Attack. N Engl J Med. 2016 Apr 7;374(14):1321-31. doi: 10.1056/NEJMoa1506930. Epub 2016 Feb 17. PMID 26886418
- [Background] Bouchi R, Terashima M, Sasahara Y, Asakawa M, Fukuda T, Takeuchi T, Nakano Y, Murakami M, Minami I, Izumiyama H, Hashimoto K, Yoshimoto T, Ogawa Y. Luseogliflozin reduces epicardial fat accumulation in patients with type 2 diabetes: a pilot study. Cardiovasc Diabetol. 2017 Mar 3;16(1):32. doi: 10.1186/s12933-017-0516-8. PMID 28253918
- [Background] Ascaso JF, Pardo S, Real JT, Lorente RI, Priego A, Carmena R. Diagnosing insulin resistance by simple quantitative methods in subjects with normal glucose metabolism. Diabetes Care. 2003 Dec;26(12):3320-5. doi: 10.2337/diacare.26.12.3320. PMID 14633821
- [Background] Bastarrika G, Broncano J, Schoepf UJ, Schwarz F, Lee YS, Abro JA, Costello P, Zwerner PL. Relationship between coronary artery disease and epicardial adipose tissue quantification at cardiac CT: comparison between automatic volumetric measurement and manual bidimensional estimation. Acad Radiol. 2010 Jun;17(6):727-34. doi: 10.1016/j.acra.2010.01.015. Epub 2010 Apr 3. PMID 20363161
- [Background] Hindso L, Jakobsen LS, Jacobsen C, Lynnerup N, Banner J. Epicardial adipose tissue volume estimation by postmortem computed tomography of eviscerated hearts. Forensic Sci Med Pathol. 2017 Dec;13(4):468-472. doi: 10.1007/s12024-017-9930-1. Epub 2017 Nov 2. PMID 29098638
- [Background] Oda S, Utsunomiya D, Funama Y, Yuki H, Kidoh M, Nakaura T, Takaoka H, Matsumura M, Katahira K, Noda K, Oshima S, Tokuyasu S, Yamashita Y. Effect of iterative reconstruction on variability and reproducibility of epicardial fat volume quantification by cardiac CT. J Cardiovasc Comput Tomogr. 2016 Mar-Apr;10(2):150-5. doi: 10.1016/j.jcct.2015.10.006. Epub 2015 Nov 3. PMID 26560351
- [Background] Ding X, Terzopoulos D, Diaz-Zamudio M, Berman DS, Slomka PJ, Dey D. Automated pericardium delineation and epicardial fat volume quantification from noncontrast CT. Med Phys. 2015 Sep;42(9):5015-26. doi: 10.1118/1.4927375. PMID 26328952
- [Background] Spearman JV, Renker M, Schoepf UJ, Krazinski AW, Herbert TL, De Cecco CN, Nietert PJ, Meinel FG. Prognostic value of epicardial fat volume measurements by computed tomography: a systematic review of the literature. Eur Radiol. 2015 Nov;25(11):3372-81. doi: 10.1007/s00330-015-3765-5. Epub 2015 Apr 30. PMID 25925354
- [Background] Iacobellis G. Local and systemic effects of the multifaceted epicardial adipose tissue depot. Nat Rev Endocrinol. 2015 Jun;11(6):363-71. doi: 10.1038/nrendo.2015.58. Epub 2015 Apr 7. PMID 25850659
- [Background] Antoniades C, Shirodaria C, Warrick N, Cai S, de Bono J, Lee J, Leeson P, Neubauer S, Ratnatunga C, Pillai R, Refsum H, Channon KM. 5-methyltetrahydrofolate rapidly improves endothelial function and decreases superoxide production in human vessels: effects on vascular tetrahydrobiopterin availability and endothelial nitric oxide synthase coupling. Circulation. 2006 Sep 12;114(11):1193-201. doi: 10.1161/CIRCULATIONAHA.106.612325. Epub 2006 Aug 28. PMID 16940192
- [Background] Margaritis M, Sanna F, Lazaros G, Akoumianakis I, Patel S, Antonopoulos AS, Duke C, Herdman L, Psarros C, Oikonomou EK, Shirodaria C, Petrou M, Sayeed R, Krasopoulos G, Lee R, Tousoulis D, Channon KM, Antoniades C. Predictive value of telomere length on outcome following acute myocardial infarction: evidence for contrasting effects of vascular vs. blood oxidative stress. Eur Heart J. 2017 Nov 1;38(41):3094-3104. doi: 10.1093/eurheartj/ehx177. PMID 28444175
- [Background] Oikonomou EK, Antoniades C. The role of adipose tissue in cardiovascular health and disease. Nat Rev Cardiol. 2019 Feb;16(2):83-99. doi: 10.1038/s41569-018-0097-6. PMID 30287946
- [Background] Antonopoulos AS, Sanna F, Sabharwal N, Thomas S, Oikonomou EK, Herdman L, Margaritis M, Shirodaria C, Kampoli AM, Akoumianakis I, Petrou M, Sayeed R, Krasopoulos G, Psarros C, Ciccone P, Brophy CM, Digby J, Kelion A, Uberoi R, Anthony S, Alexopoulos N, Tousoulis D, Achenbach S, Neubauer S, Channon KM, Antoniades C. Detecting human coronary inflammation by imaging perivascular fat. Sci Transl Med. 2017 Jul 12;9(398):eaal2658. doi: 10.1126/scitranslmed.aal2658. PMID 28701474
- [Background] Kluner LV, Oikonomou EK, Antoniades C. Assessing Cardiovascular Risk by Using the Fat Attenuation Index in Coronary CT Angiography. Radiol Cardiothorac Imaging. 2021 Feb 25;3(1):e200563. doi: 10.1148/ryct.2021200563. eCollection 2021 Feb. PMID 33778665
- [Result] Patel VB, Shah S, Verma S, Oudit GY. Epicardial adipose tissue as a metabolic transducer: role in heart failure and coronary artery disease. Heart Fail Rev. 2017 Nov;22(6):889-902. doi: 10.1007/s10741-017-9644-1. PMID 28762019

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT06557811/Prot_SAP_000.pdf